CLINICAL TRIAL: NCT07157878
Title: Gingival Crevicular Fluid Oxidized Low-Density Lipoprotein Levels in Health and Stage III/IV Periodontitis: A Cross-Sectional Comparative Study
Brief Title: Gingival Crevicular Fluid Oxidized Low-Density Lipoprotein Levels in Health and Stage III/IV Periodontitis
Acronym: LDL in GCF
Status: Not yet recruiting | Type: Observational
Sponsor: shaimaa hamdy (Other)
Responsible Party: Sponsor-Investigator, shaimaa hamdy, lecturer of periodontology, Minia University
Organization: Minia University (Other)
Other Study IDs: GCF+ advanced periodontitis; committee 1166 (Other: ethical committee faculty of dentistry minia university)
Record Dates: First submitted 2025-08-19; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Periodontal Diseases; LDL Hyperlipoproteinemia
Keywords: Periodontitis; LDL; GCF; periodontal health
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — A gingival crevicular fluid sample was taken for LDL detection to assess the correlation between periodontitis and LDL
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: periodontally healthy participants
- study group: periodontitis stage 3 and 4

SUMMARY:
Periodontitis is a chronic, multifactorial inflammatory disease primarily caused by dysbiotic plaque biofilms, characterized by the progressive destruction of the supporting structures of the teeth. In advanced stages (Stage III/IV), periodontitis leads to significant attachment and bone loss, often culminating in tooth loss and a negative impact on the patient's quality of life. Recent evidence has emphasized the systemic implications of periodontal inflammation, suggesting a bidirectional relationship between periodontitis and various systemic conditions, especially cardiovascular diseases

DETAILED DESCRIPTION:
Oxidative stress has emerged as a key pathogenic mechanism linking periodontal inflammation with systemic diseases. Among the oxidative stress-related biomarkers, oxidized low-density lipoprotein (oxLDL) has gained attention due to its pro-inflammatory, atherogenic, and cytotoxic properties. oxLDL is known to accumulate in vascular walls and contributes to the initiation and progression of atherosclerosis. Its role in periodontal disease, however, remains less well characterized. Gingival crevicular fluid (GCF) is a non-invasive biological fluid that reflects the inflammatory status of the periodontal tissues. Measuring oxLDL levels in GCF may provide valuable insight into the local oxidative burden associated with periodontal destruction. It may also help elucidate the mechanistic link between periodontal and systemic inflammatory diseases. While several studies have investigated oxLDL levels in serum in patients with periodontitis, only limited data exist regarding its levels in GCF, particularly among elderly populations who are more prone to both periodontitis and oxidative stress-related diseases. Understanding these levels could provide novel biomarkers for disease severity and progression, potentially guiding future preventive and therapeutic strategies The detection of elevated oxLDL levels in gingival crevicular fluid (GCF) could therefore serve as a meaningful, site-specific biomarker for disease activity and severity in older populations. Investigating this relationship could enhance our understanding of the oxidative mechanisms underpinning periodontal breakdown and help identify new diagnostic or prognostic markers, particularly in geriatric patients with complex medical profiles Aim of the Study To compare the levels of oxidized low-density lipoprotein (oxLDL) in gingival crevicular fluid (GCF) between healthy individuals and patients with Stage III/IV periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* For all participants (applies to both groups):

  1. Age 30-60 years.
  2. Systemically healthy (based on medical history and physician clearance, if needed).
  3. No history of periodontal treatment within the last 6 months.

Exclusion Criteria:

* 1. History of systemic diseases affecting periodontium (e.g., uncontrolled diabetes, autoimmune diseases, osteoporosis).

  2. Current or past diagnosis of Alzheimer's disease or other neurodegenerative disorders.

  3. Use of medications affecting periodontal status (e.g., immunosuppressants, long-term corticosteroids, anticonvulsants).

  4. Antibiotic or anti-inflammatory therapy within the past 3 months. 5. Current smokers or history of smoking in the past year.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cross sectional study in upper egypt to detect the level of LDL in advanced periodontitis patient
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
The concentration of oxLDL in GCF | at baseline (day1)
  The concentration of oxLDL in GCF, measured in pg/mL, in geriatric patients with Stage III/IV periodontitis compared to periodontally healthy geriatric individuals.

CONTACTS AND LOCATIONS:
Overall Officials: shaimaa Hamdy, lecturer, Study Chair — lecturer of periodontology Nahda University

IPD SHARING:
Plan to Share IPD: No
After completion of the study and complete publication, I will share all data